CLINICAL TRIAL: NCT00825318
Title: Pilot Trial To Study Blood Pressure, Weight and Hydration State in Patients Undergoing A Treatment Regimen of Daily Ultrafiltration and Twice-weekly Hemodialysis As Compared to Conventional Three Times Per Week Hemodialysis
Brief Title: Comparison Study of Daily Ultrafiltration and Twice-weekly Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renal Research Institute (Other)
Collaborators: Vizio Medical Devices (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 004-09
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: End-stage Renal Disease
Keywords: End-stage renal disease; Chronic kidney disease; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Ultrafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daily ultrafiltration (Experimental): During the treatment phase of the study, the subject will undergo ultrafiltration 6 times a week and hemodialysis 2 times a week.
  Interventions: Procedure: Ultrafiltration

INTERVENTIONS:
Procedure: Ultrafiltration — Frequency of ultrafiltration is increased from the conventional 3 times a week to 6 times a week.

SUMMARY:
In this study, the researchers want to find out how patients who have ultrafiltration (removal of excess fluid) 6 times a week and twice-weekly dialysis (removal of excess fluid and waste products) do in terms of their blood pressure and weight. The researchers believe that maintaining patients at their estimated target weight throughout the week using daily ultrafiltration will reduce their blood pressure to levels shown in other similar studies. Such a reduction in blood pressure may reduce the incidence of cerebral vascular disease, peripheral vascular disease, coronary artery disease, and congestive heart failure. The researchers also believe that patients' quality of life will improve while they are undergoing daily ultrafiltration.

Studies show that more frequent dialysis treatments result in fewer symptoms for patients. The patients feel better and avoid the weight gains and symptoms that patients have on three times a week dialysis. In addition, their blood lab results are better controlled, requiring less medication.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years and less than or equal to 80 years
* Stable three treatments per week dialysis schedule for at least three months prior to beginning the study
* Residual renal clearance <1.5ml/min per 35L of urea volume
* Pre-dialysis serum sodium levels of greater than 136 mEq/L

Exclusion Criteria:

* Non-compliance with hemodialysis treatments--defined as missing more than 1 treatment over the 3 month period prior to the study
* Unable to verbally communicate in English or Spanish
* Current requirement for hemodialysis more than three times per week due to medical comorbidity (including fourth session for ultrafiltration)
* Currently on daily or nocturnal hemodialysis, or less than 3 months since discontinued such treatment
* Expected geographic unavailability at dialysis center during any phase of the trial
* Less than 3 months since the patient returned after acute rejection resulting in allograft failure
* Currently in acute care or chronic care hospital
* Pregnancy
* Current involvement in any non-observational trial
* Unable or unwilling to follow the study protocol for any reason (including mental incompetence)
* Unable or unwilling to provide informed consent or sign IRB-approved consent form
* Pace maker, implantable pump, artificial joint
* Amputation of a limb

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan W Levin, MD, Principal Investigator — Renal Research Institute
Locations (3):
- United States (3):
  - Irving Place Dialysis Center, New York, New York
  - Upper Manhattan Dialysis Center, New York, New York
  - Yorkville Dialysis Center, New York, New York

REFERENCES:
- [Result] Bytzer P. [Laxative abuse]. Ugeskr Laeger. 1986 Jun 2;148(23):1387-9. No abstract available. Danish. PMID 3727139

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily Ultrafiltration
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Daily Ultrafiltration
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Blood Pressure
Time Frame: Prestudy Phase (retrospective analysis, 3 months), Daily Ultrafiltration Phase (4 weeks), Return Phase (4 weeks)
Measure: Mean (Full Range); unit: mm Hg
Groups:
- Prestudy Phase: During the prestudy phase, baseline 3-month retrospective data were collected for all 13 patients prior to initiation of the daily UF phase.
- Daily Ultrafiltration Phase: During the Daily UF phase of the study, the subject will undergo ultrafiltration 6 times a week and hemodialysis 2 times a week.
- Return Phase: During the Return phase, patients resumed their prior schedule of three weekly HD and UF sessions for 4 weeks. Systolic and diastolic BPs were measured before and after treatments.
Arm/Group | Prestudy Phase | Daily Ultrafiltration Phase | Return Phase
Number analyzed (Participants) | 13 | 12 | 12
mm Hg | 110 [84 to 133] | 95 [84 to 111] | 106 [92 to 121]

ADVERSE EVENTS:
Arm/Group | Prestudy Phase | Daily Ultrafiltration Phase | Return Phase
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/13 | 1/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prestudy Phase (N=0) | Daily Ultrafiltration Phase (N=13) | Return Phase (N=13)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Elevated Potassium (Metabolism and nutrition disorders) | 0 | 0 | 1 (1)
Elevated Glucose Level (Metabolism and nutrition disorders) | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes